CLINICAL TRIAL: NCT05789797
Title: Non-interventional, Prospective Study of Safety and Efficiency of the Drug Remaxol® (NTFF POLYSAN Ltd., Russia) in Patients With Drug-induced Liver Injuries During Cancer Chemotherapy.
Brief Title: Remaxol® in Patients With Drug-induced Liver Injuries During Cancer Chemotherapy
Status: Completed | Type: Observational
Sponsor: POLYSAN Scientific & Technological Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Other Study IDs: Remaxol\2022\03
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-06

CONDITIONS: Cancer; Drug Induced Liver Injury
Keywords: cancer; drug induced liver injury; remaxol
MeSH Terms: conditions — Neoplasms; Chemical and Drug Induced Liver Injury | interventions — Remaxol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- The control group: Ademethionine, lyophilisate for solution for intravenous and intramuscular injection, by intravenous drop infusion in the dose of 800 mg/day, on everyday basis for 14 days
- The test group: Remaxol®, solution for infusions, by intravenous drop infusion in the dose of 400 ml/day, on everyday basis for 12 days
  Interventions: Drug: Remaxol

INTERVENTIONS:
Drug: Remaxol — Remaxol®, solution for infusions, by intravenous drop infusion in the dose of 400 ml/day, on everyday basis for 12 days
  Groups: The test group

SUMMARY:
Cancer has moved from the tenth place to the second one over the last 100 years, being inferior to only cardiovascular diseases in morbidity and mortality.

40 % of hepatitis cases in patients older than 40 years and 25 % of cases of fulminant hepatic failure (FHF) are caused by drug hepatic toxicity. Cases of acute drug-induced hepatitis (ADIH) make 15-20 % of patients with fulminant hepatitis in Western Europe.

ELIGIBILITY:
Inclusion Criteria:

* The study can include all patients who are scheduled, at a physician's discretion, to receive the therapy with the drug Remaxol®, solution for infusions, or Ademethionine, lyophilizate for solution for intravenous and intramuscular injection, according to the approved instruction for the medical use of the drug and established clinical practice of a healthcare facility, and who meet all the following criteria:

  1. Males and females aged from 40 to 70 years inclusive.
  2. Verified diagnosis of neoplasm (morphologically proven).
  3. Receiving the course polychemotherapy (PCT).
  4. PCT regimens with pronounced hepatotoxic effects, which use drugs from the following pharmacologic classes:

     1. Competitive antagonists (5-Fluorouracil, Methotrexate etc.);
     2. Alkylating agents (Cyclophosphamide, Oxaliplatin etc.);
     3. Antitumor antibiotics (Doxorubicin, Bleomycin etc.);
     4. Drugs influencing tubulin (Trabectedin, Paclitaxel etc.);
     5. Topoisomerase inhibitors (Irinotecan, Etoposide etc.).

  <!-- -->

  1. Contraindications for the continuation of PCT at the time of a visit to a physician for its continuation, because of developed hepatotoxicity.
  2. Stage of the treatment: supporting, hepatoprotective and detoxication therapy to correct hepatotoxicity developed during PCT, to remove it and continue the chemotherapeutic treatment.
  3. A patient is scheduled to receive one of the following infusion therapies with the following regimen, as part of the routine clinical practice:
  4. It is planned to administer the drug Remaxol®, solution for infusions, by intravenous drop infusion in the dose of 400 ml/day, on everyday basis for 12 days.
  5. It is planned to administer the drug Ademethionine, lyophilisate for solution for intravenous and intramuscular injection, by intravenous drop infusion in the dose of 800 mg/day, on everyday basis for 14 days. ECOG performance status score: 1-2 inclusive (Karnofsky score: 50-80 %).
  6. Hepatotoxicity grade according to the classification of the US National Cancer Institute (NCCN, CTC) - 2 and 3.
  7. Scores by selected parameters of CTCAE (National Cancer Institute Common Toxicity Criteria for Adverse Events) scale - I and II.
  8. Patient's written consent for participation in the study according to the current legislation.

Exclusion Criteria:

1. Pregnancy, breast-feeding.
2. Mental disorders requiring psychiatric observation.
3. Chronic alcohol abuse and/or substance abuse.
4. HIV-infection, syphilis, virus hepatitis, autoimmune hepatitis, storage diseases, tuberculosis.
5. Administration of monoclonal antibodies, (multi)kinase inhibitors during the PCT session immediately preceding this study.
6. Administration of methionine-, Ademetionine-, malate- and/or succinate-containing medicines during the last month.
7. Prescription of other malate-, succinate, or methionine-containing medicines (mexidol, cytoflavin, etc.).
8. Decompensation of any severe/clinically apparent somatic diseases of the kidneys, liver, cardiovascular system, respiratory system, endocrine system, etc., as decided by the investigating physician.
9. Contraindications mentioned in the approved instructions for use of medicines applied in the study (idiosyncrasy to the product components).
10. Disease or use of medicines, which, in the doctor's opinion, can influence safety, tolerability and efficiency of the study medicines.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients with drug-induced liver injuries, during antitumor therapy
Sampling Method: Non-Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Difference of average ALT values in both of the groups, between the two timepoints: Visit 3 vs. baseline at Visit 1 (before starting therapy with the study medicines). | Baseline, up to 15 days
Difference of average ALP values in both of the groups, between the two timepoints: Visit 3 vs. baseline at Visit 1 (before starting therapy with the study medicines). | Baseline, up to 15 days

SECONDARY OUTCOMES:
Proportion of patients achieving an ECOG patient status score of 0 from the start of study (Visit1) to Visit 4, measured in both groups | Baseline, up to 28 days
  ECOG Scale of Performance Status (Eastern Cooperative Oncology Group) - 0-4 poins 0 points - The patient is fully active, able to perform everything, as before the disease.
  4 points - Disabled, completely incapable of self-care, chained to a chair or bed
Proportion of patients who resumed a PCT session (staged session after a period of study medicines administration) within 28 days of the start of hepatotoxicity correction with study medicines (Visit 1), measured in both groups. | Baseline, up to 28 days
Proportion of patients who received a staged PCT session in full (no reduction in chemotherapy doses), measured in both groups. | Baseline, up to 28 days
Proportion of patients with grade 1 of hepatotoxicity according to the CTCAE scale, by at least 3 out of 5 parameters: ALP, ALT, AST, total and direct bilirubin, GGT, from the baseline (Visit 1) to Visit 3, measured in both groups. | Baseline, up to 15 days
  Common Terminology Criteria for Adverse Events v5.0 (CTCAE)
Proportion of patients with grade 1 of hepatotoxicity according to the CTCAE scale, by at least 3 out of 5 parameters: ALP, ALT, AST, total and direct bilirubin, GGT, from the baseline (Visit 1) to Visit 4, measured in both groups. | Baseline, up to 28 days
  Common Terminology Criteria for Adverse Events v5.0 (CTCAE)
Proportion of patients with grade 4 of hepatotoxicity according to the US National Cancer Institute (CTCAE) scale, by any of the parameters from the baseline (Visit 1) to Visit 3, measured in both groups. | Baseline, up to 15 days
  Common Terminology Criteria for Adverse Events v5.0 (CTCAE)
Proportion of patients with grade 4 of hepatotoxicity according to the US National Cancer Institute (CTCAE) scale, by any of the parameters from the baseline (Visit 1) to Visit 4, measured in both groups. | Baseline, up to 28 days
  Common Terminology Criteria for Adverse Events v5.0 (CTCAE)
Difference of average total scores in A.V. Shaposhnikov hepatotoxicity scale measured in both groups between two time points: Visit 3 vs. baseline at Visit 1 (before the therapy with study medicines). | Baseline, up to 15 days
  0 degree = 0-3 points; 1 degree = 3-8 points; 2 degree = 9-14 points; 3rd degree = 15-20 points; 4 degree = 21-25 points.
ALT changes during the study period (Visit 2, 3, 4) | Baseline, up to 15 days, up to 28 days
Proportion of patients achieving 90% or more on the Karnofsky scale from the start of the study (Visit 1) to Visit 3, measured in both groups. | Baseline, up to 15 days
  the Karnofsky score: 100% - Normal condition, no complaints 90% - Capable of normal activities, minor symptoms or signs of disease 80% - Normal activity with effort, minor symptoms or signs of disease 70% Self-supporting, incapable of normal activities or active work 60% - Sometimes needs help, but is able to satisfy most of his needs. 50% - Needs significant assistance and medical care 40% - Disabled, needs special assistance, including medical 30% - Severe disability, hospitalization is indicated, although death is not directly threatened 20% - Severe patient. Hospitalization and active treatment required 10% - Dying
Proportion of patients with full normalisation of ALT, AST by 2, 3, 4 Visits, measured in both groups. | Baseline, up to 7 days, up to 15 days, up to 28 days
Proportion of patients with full normalisation of ALP by 2, 3, 4 Visits, measured in both groups. | Baseline, up to 7 days, up to 15 days, up to 28 days
Proportion of patients with full normalisation of GGT by 2, 3, 4 Visits, measured in both groups. | Baseline, up to 7 days, up to 15 days, up to 28 days
Proportion of patients with full normalisation of total and direct bilirubin by 2, 3, 4 Visits, measured in both groups. | Baseline, up to 7 days, up to 15 days, up to 28 days
Changes in the patient's condition according to the Karnofsky score during the study (Visits 2, 3, 4) compared to the study initiation (Visit 1), expressed as a % of the baseline | Baseline, up to 7 days, up to 15 days, up to 28 days
  the Karnofsky score: 100% - Normal condition, no complaints 90% - Capable of normal activities, minor symptoms or signs of disease 80% - Normal activity with effort, minor symptoms or signs of disease 70% Self-supporting, incapable of normal activities or active work 60% - Sometimes needs help, but is able to satisfy most of his needs. 50% - Needs significant assistance and medical care 40% - Disabled, needs special assistance, including medical 30% - Severe disability, hospitalization is indicated, although death is not directly threatened 20% - Severe patient. Hospitalization and active treatment required 10% - Dying
Changes in the patient's condition according to the ECOG Scale, during the study period (Visits 2, 3, 4) as compared to the study initiation (Visit 1), expressed as a score and as a % of the baseline | Baseline, up to 7 days, up to 15 days, up to 28 days
  ECOG Scale of Performance Status (Eastern Cooperative Oncology Group) - 0-4 poins 0 points - The patient is fully active, able to perform everything, as before the disease.
  4 points - Disabled, completely incapable of self-care, chained to a chair or bed
Proportion of patients with detected toxic damage to at least one system or organ (by selected parameters), according to the criteria of common toxicity grade III of the CTCAE scale, from the baseline (Visit 1) to Visit 3, measured in both groups. | Baseline, up to 15 days
  Common Terminology Criteria for Adverse Events v5.0 (CTCAE)
Proportion of patients with detected toxic damage to at least one system or organ (by selected parameters), according to the criteria of common toxicity grade III of the CTCAE scale, from the baseline (Visit 1) to Visit 4, measured in both groups. | Baseline, up to 28 days
  Common Terminology Criteria for Adverse Events v5.0 (CTCAE)

CONTACTS AND LOCATIONS:
Locations (5):
- Russia (5):
  - State Budget-Funded Health Institution Kryzhanovsky Krasnoyarsk Krai Clinical Cancer Centre, Krasnoyarsk
  - North-West Center of Evidence-Based Medicine, Saint Petersburg
  - Pirogov Clinic of High Medical Technologies, St. Petersburg State University, Saint Petersburg
  - St. Petersburg State Budget-Funded Health Institution City Clinical Cancer Centre, Saint Petersburg
  - Republican Clinical Cancer Centre, Ufa

IPD SHARING:
Plan to Share IPD: No